CLINICAL TRIAL: NCT01340040
Title: A Phase 1, Open-label, Single-arm, Dose-escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI-573, a Fully Human Monoclonal Antibody Directed Against Insulin-like Growth Factors I and II, in Japanese Subjects With Advanced Solid Tumours Refractory to Standard Therapy or for Which No Standard Therapy Exists
Brief Title: Dose-escalation Study to Assess Safety, Tolerability and Pharmacokinetics of MEDI-573 in Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5621C00006
Record Dates: First submitted 2011-04-11; First posted 2011-04-21 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Cancer; Advanced Solid Malignancies
Keywords: Phase I; cancer; solid tumours; advanced solid malignancies; dose escalation; Insulin like growth factor; Japanese
MeSH Terms: conditions — Neoplasms | interventions — dusigitumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEDI-573 (Experimental): MEDI-573
  Interventions: Drug: MEDI-573

INTERVENTIONS:
Drug: MEDI-573 — MEDI-573 will be administrated once 7 days in Cohort 1 and 2, and once every 21 days in Cohort 3 as a IV infusion as part of a 21-day treatment cycle.

SUMMARY:
The primary purpose of this study is to explore the safety and tolerability of MEDI-573 in Japanese subjects with advanced solid tumours refractory to standard therapy or for which no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Japanese men or women at least 20 years of age
* Histological or cytological confirmation of a solid, malignant tumour excluding lymphoma that is refractory to standard therapies or for which no standard therapies exist
* WHO performance status 0-2 with no deterioration over the previous 2 weeks

Exclusion Criteria:

* Previous therapy with medication against IGF (ie, monoclonal antibodies with IGF-1R or IGF-targeting tyrosine kinase inhibitors)
* Inadequate bone marrow reserve or organ function
* Poorly controlled diabetes mellitus as defined by the investigator's assessment and/or glycosylated hemoglobin (HbA1c) reading > 6.5% within 28 days prior to the first dose of MEDI-573
* History of allergy or reaction to any component of the MEDI-573 formulation or drugs with a similar chemical structure or class to MEDI-573

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (based on CTCAE version 4.0), laboratory values, vital sign measurements, ECG, Physical Examination | All AEs will be collected throughout the study, from informed consent until 30 days after the end of study treatment.
  The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.

SECONDARY OUTCOMES:
Immunogenicity of MEDI-573 (by measuring anti-MEDI-573 antibodies) | For Cohorts 1, 2 and 3:day 1 (pre-dose) of every cycle; 30 days after the last dose; 3 months after the last dose
  The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.
Anti-tumor activity of MEDI-573 using Response Evaluation Criteria in Solid Tumors(RECIST) | Tumor assessment by RECIST 1.1 every 2 cycles
  subjects who discontinue the study treatment for reasons other than disease progression or initiation of alternative anticancer therapy will undergo tumor assessment 3 months after the last dose of MEDI-573). The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.
Pharmacokinetics, - Cmax | For Cohorts 1, 2 and 3:Multiple timepoints taken, begining at Day 1 and until 30 days after last dose.
  The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.
Pharmacokinetics,- Cmax at steady state (Cmax, ss) | For Cohorts 1, 2 and 3: Multiple timepoints taken, begining at Day 1 and until 30 days after last dose.
  The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.
Pharmacokinetics - time to maximum concentration (tmax) | For Cohorts 1, 2 and 3: Multiple timepoints taken, begining at Day 1 and until 30 days after last dose.
  The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.
Pharmacokinetics, - terminal elimination rate constant (λz) | For Cohorts 1, 2 and 3: Multiple timepoints taken, begining at Day 1 and until 30 days after last dose.
  The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.
Pharmacokinetics - (AUC(0-t)) | For Cohorts 1, 2 and 3: Multiple timepoints taken, begining at Day 1 and until 30 days after last dose.
  The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.
Pharmacokinetics - total clearance and terminal phase (Vz) of MEDI-573 | For Cohorts 1, 2 and 3: Multiple timepoints taken, begining at Day 1 and until 30 days after last dose.
  The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.
Pharmacodynamics: - Insulin-like growth factor (IGF)-I and IGF-II on circulating plasma levels of MEDI-573 | For Cohorts 1, 2 and 3: Multiple timepoints taken, begining at Day 1 and until 30 days after last dose.
  The total duration of this time frame can not be specified, as it depends on the number of treatments the subject may receive.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Bradley, MD, Study Director — MedImmune LLC
Locations (1):
- Research Site, Matsuyama, Ehime, Japan

REFERENCES:
- [Derived] Iguchi H, Nishina T, Nogami N, Kozuki T, Yamagiwa Y, Yagawa K. Phase I dose-escalation study evaluating safety, tolerability and pharmacokinetics of MEDI-573, a dual IGF-I/II neutralizing antibody, in Japanese patients with advanced solid tumours. Invest New Drugs. 2015 Feb;33(1):194-200. doi: 10.1007/s10637-014-0170-x. Epub 2014 Oct 25. PMID 25342141
- See also: Protocol Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=512&filename=MEDI-573_D5621C00006_Protocol_Redacted_final.pdf